CLINICAL TRIAL: NCT00191438
Title: Phase III Study of Docetaxel in Combination With Gemcitabine Versus Docetaxel in Combination With Capecitabine in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase III Study of Gemcitabine Plus a Cytotoxic Agent Versus Two Cytotoxic Agents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6136; B9E-MC-S273
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Capecitabine; Docetaxel

INTERVENTIONS:
Drug: gemcitabine
Drug: capecitabine
Drug: docetaxel

SUMMARY:
This is a phase III randomized study which compares two different regimens of chemotherapy. The purpose of the study is to determine which of the two regimens will make the tumor smaller or disappear, and for how long. In addition the disease-related symptoms will be evaluated. The safety of the drugs will be determined based upon evaluation of the side effects

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced and/or metastatic breast cancer.
* Measurable disease
* Previously treated with anthracycline

Exclusion Criteria:

* Patients with inflammatory breast disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-10; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival. The final analysis will occur when 250 patients have progressed or died.

SECONDARY OUTCOMES:
Overall toxicity
Quality of Life
Overall Survival
Overall Response Rate
Time to Treatment Failure

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon-Fri 9AM-5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem, Netherlands
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia, Valencia, Spain
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com